CLINICAL TRIAL: NCT02451670
Title: Reducing Cardiovascular Risk in Adults With Serious Mental Illness Using an Electronic Medical Record-based Clinical Decision Support
Brief Title: Reducing Cardiovascular Risk in Adults With Serious Mental Illness
Acronym: SMIWizard
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Essentia Health (Other); National Institute of Mental Health (NIMH) (NIH); Park Nicollet Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A13-154; U19MH092201 (NIH)
Record Dates: First submitted 2015-05-18; First posted 2015-05-22 (Estimated); Results first posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-03

CONDITIONS: Chronic Disease; Mental Disorder; Health Behavior; Bipolar Disorder; Schizophrenia
MeSH Terms: conditions — Chronic Disease; Mental Disorders; Health Behavior; Bipolar Disorder; Schizophrenia

STUDY DESIGN:
Intervention Model Description: Clinics have been randomized into a treatment and a control arm.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prioritized Clinical Decision Support (Experimental): Patients receiving care in clinics randomized to the intervention arm of the study and their primary care providers were presented with patient-specific written advice as to prioritized treatment and lifestyle changes that could reduce their cardiovascular risk, prompted by an electronic health record-based alert during their primary care visit.
  Interventions: Behavioral: Prioritized Clinical Decision Support
- Usual Care (No Intervention): Patients receiving care in clinics randomized to the usual care arm of the study and their providers were not presented with the prioritized clinical decision support.

INTERVENTIONS:
Behavioral: Prioritized Clinical Decision Support — After entry of blood pressure data at all primary care visits, relevant electronic health record data were automatically extracted, encrypted and processed through Web-based clinical algorithms that determined if the patient met intervention eligibility criteria. In intervention clinics, the rooming staff received a best practice alert and printed patient and primary care provider versions of the clinical decision support that identified evidence-based treatment options for any uncontrolled cardiovascular risk factors and prioritized treatment recommendations based on potential cardiovascular risk reduction. Cardiovascular risk factors addressed in study participants were control of lipids, blood pressure, weight, tobacco, glucose and appropriate aspirin use. In control clinics, rooming staff did not receive a best practice alert and patients and primary care providers did not receive and were not able to access the clinical decision support.
  Arms: Prioritized Clinical Decision Support

SUMMARY:
This purpose of this study is to adapt, implement and test the ability of a sophisticated point-of-care electronic health record-based clinical decision support that identifies and prioritizes all available evidence-based treatment options to reduce cardiovascular risk in patients with serious mental illness.

DETAILED DESCRIPTION:
This study adapted a point-of-care electronic health record-based clinical decision support system (The Cardiovascular Wizard) to help primary care providers identify, provide appropriate care for, and control cardiovascular risk factors for patients with serious mental illness (bipolar disorder, schizophrenia, schizo-affective disorder). The Cardiovascular Wizard is designed to educate primary care providers about the increased risk of cardiovascular disease and mortality in people with serious mental illness, identify elevated cardiovascular risk factors in patients with serious mental illness, identify elevated cardiovascular risk factors in patients with serious mental illness, prioritize these cardiovascular risk based on how much improvement in cardiovascular risk a patient would experience if the cardiovascular risk factor was adequately addressed, recommend specific medications and other interventions to decrease each elevated cardiovascular risk factor, and provide this information in an easy-to-understand format for both patients with serious mental illness and their primary care providers.

The Cardiovascular Wizard was printed in intervention clinics and (i) compiled lab data (most recent glycated hemoglobin, systolic blood pressure and low-density lipoprotein levels), body mass index, smoking status, and aspirin use, (ii) calculated a modifiable 10 year cardiovascular risk for stroke or heart attack using the American College of Cardiology/American Heart Association 10-year atherosclerotic cardiovascular disease risk equation, (iii) prioritized clinical domains based on the absolute risk reduction for each component, (iv) compiled information related to liver and renal function, creatinine kinase level, and previous diagnoses (Congestive Heart Failure, Cardiovascular Disease, Diabetes Mellitus, and (v) provided recommendations for intensification of therapy for glycated hemoglobin, systolic blood pressure, and/or low-density lipoproteins if not at goal. Recommendations were based on evidence-based protocols including Joint National Committee, American Diabetes Association, and the Institute for Clinical Systems Improvement.

ELIGIBILITY:
Inclusion Criteria:

* Serious Mental Illness diagnosis
* Age 18-75
* Index visit during the enrollment period
* First primary care visit where patient was not at goal for at least one of the six cardiovascular risk factor areas, and patient was not pregnant
* One or more post-index visits during the intervention period

Exclusion Criteria:

* No Serious Mental Illness diagnosis
* Under age 18 or over age 75
* In hospice or nursing home
* At goal for all cardiovascular risk 6 areas
* On research exclusion list

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10347 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca C Rossom, MD, Principal Investigator — HealthPartners Institute
Locations (3):
- United States (3):
  - Essentia Health, Duluth, Minnesota
  - Park Nicollet Clinic, Minneapolis, Minnesota
  - HealthPartners, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weiner M, Warren L, Fiedorowicz JG. Cardiovascular morbidity and mortality in bipolar disorder. Ann Clin Psychiatry. 2011 Feb;23(1):40-7. PMID 21318195
- [Background] Osborn DP, Levy G, Nazareth I, Petersen I, Islam A, King MB. Relative risk of cardiovascular and cancer mortality in people with severe mental illness from the United Kingdom's General Practice Rsearch Database. Arch Gen Psychiatry. 2007 Feb;64(2):242-9. doi: 10.1001/archpsyc.64.2.242. PMID 17283292
- [Background] De Hert M, Dekker JM, Wood D, Kahl KG, Holt RI, Moller HJ. Cardiovascular disease and diabetes in people with severe mental illness position statement from the European Psychiatric Association (EPA), supported by the European Association for the Study of Diabetes (EASD) and the European Society of Cardiology (ESC). Eur Psychiatry. 2009 Sep;24(6):412-24. doi: 10.1016/j.eurpsy.2009.01.005. Epub 2009 Aug 13. PMID 19682863
- [Background] O'Connor PJ, Crain AL, Rush WA, Sperl-Hillen JM, Gutenkauf JJ, Duncan JE. Impact of an electronic medical record on diabetes quality of care. Ann Fam Med. 2005 Jul-Aug;3(4):300-6. doi: 10.1370/afm.327. PMID 16046561
- [Background] Osby U, Correia N, Brandt L, Ekbom A, Sparen P. Mortality and causes of death in schizophrenia in Stockholm county, Sweden. Schizophr Res. 2000 Sep 29;45(1-2):21-8. doi: 10.1016/s0920-9964(99)00191-7. PMID 10978869
- [Background] Hennekens CH, Hennekens AR, Hollar D, Casey DE. Schizophrenia and increased risks of cardiovascular disease. Am Heart J. 2005 Dec;150(6):1115-21. doi: 10.1016/j.ahj.2005.02.007. PMID 16338246
- [Background] Dixon L, Postrado L, Delahanty J, Fischer PJ, Lehman A. The association of medical comorbidity in schizophrenia with poor physical and mental health. J Nerv Ment Dis. 1999 Aug;187(8):496-502. doi: 10.1097/00005053-199908000-00006. PMID 10463067
- [Background] Davidson S, Judd F, Jolley D, Hocking B, Thompson S, Hyland B. Cardiovascular risk factors for people with mental illness. Aust N Z J Psychiatry. 2001 Apr;35(2):196-202. doi: 10.1046/j.1440-1614.2001.00877.x. PMID 11284901
- [Background] Druss BG, Bradford WD, Rosenheck RA, Radford MJ, Krumholz HM. Quality of medical care and excess mortality in older patients with mental disorders. Arch Gen Psychiatry. 2001 Jun;58(6):565-72. doi: 10.1001/archpsyc.58.6.565. PMID 11386985
- [Background] Trangle M, Gary M, Paul G, Christensen R. Minnesota 10 by 10. Reducing morbidity and mortality in people with serious mental illnesses. Minn Med. 2010 Jun;93(6):38-41. PMID 20827954
- [Background] Goff DC, Sullivan LM, McEvoy JP, Meyer JM, Nasrallah HA, Daumit GL, Lamberti S, D'Agostino RB, Stroup TS, Davis S, Lieberman JA. A comparison of ten-year cardiac risk estimates in schizophrenia patients from the CATIE study and matched controls. Schizophr Res. 2005 Dec 1;80(1):45-53. doi: 10.1016/j.schres.2005.08.010. Epub 2005 Sep 28. PMID 16198088
- [Background] Newcomer JW. Medical risk in patients with bipolar disorder and schizophrenia. J Clin Psychiatry. 2006;67 Suppl 9:25-30; discussion 36-42. PMID 16965186
- [Background] Kilbourne AM, Cornelius JR, Han X, Pincus HA, Shad M, Salloum I, Conigliaro J, Haas GL. Burden of general medical conditions among individuals with bipolar disorder. Bipolar Disord. 2004 Oct;6(5):368-73. doi: 10.1111/j.1399-5618.2004.00138.x. PMID 15383128
- [Background] Birkenaes AB, Opjordsmoen S, Brunborg C, Engh JA, Jonsdottir H, Ringen PA, Simonsen C, Vaskinn A, Birkeland KI, Friis S, Sundet K, Andreassen OA. The level of cardiovascular risk factors in bipolar disorder equals that of schizophrenia: a comparative study. J Clin Psychiatry. 2007 Jun;68(6):917-23. doi: 10.4088/jcp.v68n0614. PMID 17592917
- [Background] Wong CK, Tang EW, Herbison P, Birmingham B, Barclay L, Fu SY. Pre-existent depression in the 2 weeks before an acute coronary syndrome can be associated with delayed presentation of the heart attack. QJM. 2008 Feb;101(2):137-44. doi: 10.1093/qjmed/hcm153. Epub 2008 Jan 10. PMID 18187481
- [Background] Druss BG. Improving medical care for persons with serious mental illness: challenges and solutions. J Clin Psychiatry. 2007;68 Suppl 4:40-4. PMID 17539699
- [Background] Laursen TM, Munk-Olsen T, Agerbo E, Gasse C, Mortensen PB. Somatic hospital contacts, invasive cardiac procedures, and mortality from heart disease in patients with severe mental disorder. Arch Gen Psychiatry. 2009 Jul;66(7):713-20. doi: 10.1001/archgenpsychiatry.2009.61. PMID 19581562
- [Background] Mackin P, Bishop DR, Watkinson HM. A prospective study of monitoring practices for metabolic disease in antipsychotic-treated community psychiatric patients. BMC Psychiatry. 2007 Jun 25;7:28. doi: 10.1186/1471-244X-7-28. PMID 17592636
- [Background] Shah SU, White A, White S, Littler WA. Heart and mind: (1) relationship between cardiovascular and psychiatric conditions. Postgrad Med J. 2004 Dec;80(950):683-9. doi: 10.1136/pgmj.2003.014662. PMID 15579605
- [Background] Sowden GL, Huffman JC. The impact of mental illness on cardiac outcomes: a review for the cardiologist. Int J Cardiol. 2009 Feb 6;132(1):30-7. doi: 10.1016/j.ijcard.2008.10.002. Epub 2008 Nov 11. PMID 19004512
- [Background] Taylor V, MacQueen G. Associations between bipolar disorder and metabolic syndrome: A review. J Clin Psychiatry. 2006 Jul;67(7):1034-41. doi: 10.4088/jcp.v67n0704. PMID 16889445
- [Background] Klumpers UM, Boom K, Janssen FM, Tulen JH, Loonen AJ. Cardiovascular risk factors in outpatients with bipolar disorder. Pharmacopsychiatry. 2004 Sep;37(5):211-6. doi: 10.1055/s-2004-832594. PMID 15470799
- [Background] American Diabetes Association; American Psychiatric Association; American Association of Clinical Endocrinologists; North American Association for the Study of Obesity. Consensus development conference on antipsychotic drugs and obesity and diabetes. Diabetes Care. 2004 Feb;27(2):596-601. doi: 10.2337/diacare.27.2.596. No abstract available. PMID 14747245
- [Background] Druss BG, Bradford DW, Rosenheck RA, Radford MJ, Krumholz HM. Mental disorders and use of cardiovascular procedures after myocardial infarction. JAMA. 2000 Jan 26;283(4):506-11. doi: 10.1001/jama.283.4.506. PMID 10659877
- [Background] Frayne SM, Halanych JH, Miller DR, Wang F, Lin H, Pogach L, Sharkansky EJ, Keane TM, Skinner KM, Rosen CS, Berlowitz DR. Disparities in diabetes care: impact of mental illness. Arch Intern Med. 2005 Dec 12-26;165(22):2631-8. doi: 10.1001/archinte.165.22.2631. PMID 16344421
- [Background] Desai MM, Rosenheck RA, Druss BG, Perlin JB. Mental disorders and quality of diabetes care in the veterans health administration. Am J Psychiatry. 2002 Sep;159(9):1584-90. doi: 10.1176/appi.ajp.159.9.1584. PMID 12202281
- [Background] Fagiolini A, Chengappa KN, Soreca I, Chang J. Bipolar disorder and the metabolic syndrome: causal factors, psychiatric outcomes and economic burden. CNS Drugs. 2008;22(8):655-69. doi: 10.2165/00023210-200822080-00004. PMID 18601304
- [Background] Mitchell JE, Mackenzie TB. Cardiac effects of lithium therapy in man: a review. J Clin Psychiatry. 1982 Feb;43(2):47-51. PMID 7056703
- [Background] Glassman AH, Bigger JT Jr. Antipsychotic drugs: prolonged QTc interval, torsade de pointes, and sudden death. Am J Psychiatry. 2001 Nov;158(11):1774-82. doi: 10.1176/appi.ajp.158.11.1774. PMID 11691681
- [Background] Morriss R, Mohammed FA. Metabolism, lifestyle and bipolar affective disorder. J Psychopharmacol. 2005 Nov;19(6 Suppl):94-101. doi: 10.1177/0269881105058678. PMID 16280342
- [Background] Angst F, Stassen HH, Clayton PJ, Angst J. Mortality of patients with mood disorders: follow-up over 34-38 years. J Affect Disord. 2002 Apr;68(2-3):167-81. doi: 10.1016/s0165-0327(01)00377-9. PMID 12063145
- [Background] Ryan MC, Thakore JH. Physical consequences of schizophrenia and its treatment: the metabolic syndrome. Life Sci. 2002 Jun 7;71(3):239-57. doi: 10.1016/s0024-3205(02)01646-6. PMID 12034344
- [Background] Lieberman JA, Stroup TS, McEvoy JP, Swartz MS, Rosenheck RA, Perkins DO, Keefe RS, Davis SM, Davis CE, Lebowitz BD, Severe J, Hsiao JK; Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) Investigators. Effectiveness of antipsychotic drugs in patients with chronic schizophrenia. N Engl J Med. 2005 Sep 22;353(12):1209-23. doi: 10.1056/NEJMoa051688. Epub 2005 Sep 19. PMID 16172203
- [Background] Elmer PJ, Obarzanek E, Vollmer WM, Simons-Morton D, Stevens VJ, Young DR, Lin PH, Champagne C, Harsha DW, Svetkey LP, Ard J, Brantley PJ, Proschan MA, Erlinger TP, Appel LJ; PREMIER Collaborative Research Group. Effects of comprehensive lifestyle modification on diet, weight, physical fitness, and blood pressure control: 18-month results of a randomized trial. Ann Intern Med. 2006 Apr 4;144(7):485-95. doi: 10.7326/0003-4819-144-7-200604040-00007. PMID 16585662
- [Background] Whelton PK, Appel LJ, Espeland MA, Applegate WB, Ettinger WH Jr, Kostis JB, Kumanyika S, Lacy CR, Johnson KC, Folmar S, Cutler JA. Sodium reduction and weight loss in the treatment of hypertension in older persons: a randomized controlled trial of nonpharmacologic interventions in the elderly (TONE). TONE Collaborative Research Group. JAMA. 1998 Mar 18;279(11):839-46. doi: 10.1001/jama.279.11.839. PMID 9515998
- [Background] Daumit GL, Dickerson FB, Wang NY, Dalcin A, Jerome GJ, Anderson CA, Young DR, Frick KD, Yu A, Gennusa JV 3rd, Oefinger M, Crum RM, Charleston J, Casagrande SS, Guallar E, Goldberg RW, Campbell LM, Appel LJ. A behavioral weight-loss intervention in persons with serious mental illness. N Engl J Med. 2013 Apr 25;368(17):1594-602. doi: 10.1056/NEJMoa1214530. Epub 2013 Mar 21. PMID 23517118
- [Background] Pylvanen V, Knip M, Pakarinen A, Kotila M, Turkka J, Isojarvi JI. Serum insulin and leptin levels in valproate-associated obesity. Epilepsia. 2002 May;43(5):514-7. doi: 10.1046/j.1528-1157.2002.31501.x. PMID 12027912
- [Background] Sachs G, Bowden C, Calabrese JR, Ketter T, Thompson T, White R, Bentley B. Effects of lamotrigine and lithium on body weight during maintenance treatment of bipolar I disorder. Bipolar Disord. 2006 Apr;8(2):175-81. doi: 10.1111/j.1399-5618.2006.00308.x. PMID 16542188
- [Background] Allison DB, Mentore JL, Heo M, Chandler LP, Cappelleri JC, Infante MC, Weiden PJ. Antipsychotic-induced weight gain: a comprehensive research synthesis. Am J Psychiatry. 1999 Nov;156(11):1686-96. doi: 10.1176/ajp.156.11.1686. PMID 10553730
- [Background] Komossa K, Rummel-Kluge C, Schmid F, Hunger H, Schwarz S, El-Sayeh HG, Kissling W, Leucht S. Aripiprazole versus other atypical antipsychotics for schizophrenia. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD006569. doi: 10.1002/14651858.CD006569.pub3. PMID 19821375
- [Background] Patel JK, Buckley PF, Woolson S, Hamer RM, McEvoy JP, Perkins DO, Lieberman JA; CAFE Investigators. Metabolic profiles of second-generation antipsychotics in early psychosis: findings from the CAFE study. Schizophr Res. 2009 Jun;111(1-3):9-16. doi: 10.1016/j.schres.2009.03.025. Epub 2009 Apr 26. PMID 19398192
- [Background] Sittig DF, Wright A, Osheroff JA, Middleton B, Teich JM, Ash JS, Campbell E, Bates DW. Grand challenges in clinical decision support. J Biomed Inform. 2008 Apr;41(2):387-92. doi: 10.1016/j.jbi.2007.09.003. Epub 2007 Sep 21. PMID 18029232
- [Background] O'Connor PJ, Sperl-Hillen JM, Rush WA, Johnson PE, Amundson GH, Asche SE, Ekstrom HL, Gilmer TP. Impact of electronic health record clinical decision support on diabetes care: a randomized trial. Ann Fam Med. 2011 Jan-Feb;9(1):12-21. doi: 10.1370/afm.1196. PMID 21242556
- [Background] Leibson C, Owens T, O'Brien P, Waring S, Tangalos E, Hanson V, Plevak M, Kokmen E. Use of physician and acute care services by persons with and without Alzheimer's disease: a population-based comparison. J Am Geriatr Soc. 1999 Jul;47(7):864-9. doi: 10.1111/j.1532-5415.1999.tb03846.x. PMID 10404933
- [Background] O'Connor PJ, Desai JR, Butler JC, Kharbanda EO, Sperl-Hillen JM. Current status and future prospects for electronic point-of-care clinical decision support in diabetes care. Curr Diab Rep. 2013 Apr;13(2):172-6. doi: 10.1007/s11892-012-0350-z. PMID 23225213
- [Background] O'Connor PJ, Quiter ES, Rush WA, Wiest M, Meland JT, Ryu S. Impact of hypertension guideline implementation on blood pressure control and drug use in primary care clinics. Jt Comm J Qual Improv. 1999 Feb;25(2):68-77. doi: 10.1016/s1070-3241(16)30428-x. PMID 10027112
- [Background] Boyle RG, O'Connor PJ, Pronk NP, Tan A. Stages of change for physical activity, diet, and smoking among HMO members with chronic conditions. Am J Health Promot. 1998 Jan-Feb;12(3):170-5. doi: 10.4278/0890-1171-12.3.170. PMID 10176091
- [Background] O'Connor PJ, Asche SE, Crain AL, Rush WA, Whitebird RR, Solberg LI, Sperl-Hillen JM. Is patient readiness to change a predictor of improved glycemic control? Diabetes Care. 2004 Oct;27(10):2325-9. doi: 10.2337/diacare.27.10.2325. PMID 15451895
- [Background] O'Connor PJ, Sperl-Hillen J. Clinical and public health implications of glycemic relapse in type 2 diabetes. Nat Clin Pract Endocrinol Metab. 2007 Jan;3(1):10-1. doi: 10.1038/ncpendmet0354. No abstract available. PMID 17179924
- [Background] O'Connor PJ, Rush WA, Prochaska JO, Pronk NP, Boyle RG. Professional advice and readiness to change behavioral risk factors among members of a managed care organization. Am J Manag Care. 2001 Feb;7(2):125-30. PMID 11216330
- [Background] O'Connor PJ. Electronic medical records and diabetes care improvement: are we waiting for Godot? Diabetes Care. 2003 Mar;26(3):942-3. doi: 10.2337/diacare.26.3.942. No abstract available. PMID 12610062
- [Derived] Rossom RC, Crain AL, Waring S, Sperl-Hillen JM, Hooker SA, Miley K, O'Connor PJ. Differential Effects of an Intervention to Reduce Cardiovascular Risk for Patients With Bipolar Disorder, Schizoaffective Disorder, or Schizophrenia: A Randomized Clinical Trial. J Clin Psychiatry. 2023 Jul 5;84(4):22m14710. doi: 10.4088/JCP.22m14710. PMID 37428030
- [Derived] Sperl-Hillen JM, Anderson JP, Margolis KL, Rossom RC, Kopski KM, Averbeck BM, Rosner JA, Ekstrom HL, Dehmer SP, O'Connor PJ. Bolstering the Business Case for Adoption of Shared Decision-Making Systems in Primary Care: Randomized Controlled Trial. JMIR Form Res. 2022 Oct 6;6(10):e32666. doi: 10.2196/32666. PMID 36201392
- [Derived] Rossom RC, Hooker SA, O'Connor PJ, Crain AL, Sperl-Hillen JM. Cardiovascular Risk for Patients With and Without Schizophrenia, Schizoaffective Disorder, or Bipolar Disorder. J Am Heart Assoc. 2022 Mar 15;11(6):e021444. doi: 10.1161/JAHA.121.021444. Epub 2022 Mar 9. PMID 35261265
- [Derived] Rossom RC, Crain AL, O'Connor PJ, Waring SC, Hooker SA, Ohnsorg K, Taran A, Kopski KM, Sperl-Hillen JM. Effect of Clinical Decision Support on Cardiovascular Risk Among Adults With Bipolar Disorder, Schizoaffective Disorder, or Schizophrenia: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2022 Mar 1;5(3):e220202. doi: 10.1001/jamanetworkopen.2022.0202. PMID 35254433
- [Derived] Rossom RC, O'Connor PJ, Crain AL, Waring S, Ohnsorg K, Taran A, Kopski K, Sperl-Hillen JM. Pragmatic trial design of an intervention to reduce cardiovascular risk in people with serious mental illness. Contemp Clin Trials. 2020 Apr;91:105964. doi: 10.1016/j.cct.2020.105964. Epub 2020 Feb 20. PMID 32087336

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients with an adult primary care visit with a primary care provider in a randomized clinic were assessed for study eligibility. After entry of blood pressure data, relevant health record data were automatically extracted, encrypted and processed through Web-based clinical algorithms that determined eligibility.
Units Other Than Participants: Clinics
Groups:
- Prioritized Clinical Support: Patients and their primary care providers in the intervention arm were presented with patient-specific written advice as to prioritized treatment and lifestyle changes that could reduce their cardiovascular risk, prompted by an electronic health record-based alert during their primary care visit.
- Usual Care: Patients and their primary care providers in the usual care arm were not presented with prioritized clinical decision support.
Period: Overall Study
Arm/Group | Prioritized Clinical Support | Usual Care
Started | 5264; 47 Clinics | 5083; 38 Clinics
Completed | 4550; 47 Clinics | 4387; 38 Clinics
Not Completed | 714; 0 Clinics | 696; 0 Clinics
Not completed — Did not have qualifying follow-up visit. | 714 | 696

BASELINE CHARACTERISTICS:
Population: Patients whose data was included in the baseline analysis population met eligibility criteria, had an index visit at a randomized clinic at which they were eligible for the CV Wizard intervention, and had at least one follow-up visit in a randomized primary care clinic.
Groups:
- Prioritized Clinical Decision Support: Patients and their primary care providers were presented with patient-specific written instructions as to prioritized treatment and lifestyle changes that could reduce cardiovascular risk, prompted by an electronic health record-based alert during their primary care visits.
- Usual Care: Patients and their providers were not presented with the prioritized clinical decision support.
- Total: Total of all reporting groups
Arm/Group | Prioritized Clinical Decision Support | Usual Care | Total
Number analyzed (Participants) | 4550 | 4387 | 8937
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (13.3) | 48.1 (13.4) | 48.4 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2530 | 2393 | 4923
  Male | 2020 | 1994 | 4014
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 66 | 108
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 4508 | 4321 | 8829
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 113 | 68 | 181
  Asian | 76 | 54 | 130
  Native Hawaiian or Other Pacific Islander | 5 | 5 | 10
  Black or African American | 517 | 390 | 907
  White | 3749 | 3741 | 7490
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 90 | 129 | 219
Region of Enrollment [Number; unit: participants]
  United States | 4550 | 4387 | 8937
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 124.4 (16.6) | 124.2 (16.5) | 124.3 (16.6)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 78.3 (11.4) | 78.3 (11.4) | 78.3 (11.4)
Active Smoker [Count of Participants; unit: Participants] | 2131 | 2027 | 4158
Aspirin Use [Count of Participants; unit: Participants] — Population: Only patients that met criteria for aspirin therapy were included in this measure.
  Participants
    number analyzed (Participants) | 907 | 822 | 1729
    (all) | 519 | 461 | 980
Low-Density Lipoprotein Cholesterol [Mean (Standard Deviation); unit: mg/dl] — Population: Only patients that had a recent Low-Density Lipoprotein result in their electronic medical record were included in this measure.
  mg/dl
    number analyzed (Participants) | 3680 | 3536 | 7216
    (all) | 104.9 (35.4) | 104.6 (35.6) | 104.8 (7978)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Only patients with a recent weight in their electronic medical record were included in this measure.
  kg/m^2
    number analyzed (Participants) | 4135 | 3943 | 8078
    (all) | 32.5 (7.8) | 32.7 (7.9) | 32.6 (7.9)

OUTCOME MEASURES:

1. Primary Outcome: Predicted Annual Rate of Change in 10 Year Risk of Fatal or Nonfatal Heart Attack or Stroke
Description: A modifiable risk component for each cardiovascular risk factor not at optimal goal at the time of each encounter was calculated as the difference between total 10-year atherosclerotic cardiovascular disease risk with the patient's actual values and the goal value. Total modifiable cardiovascular risk was calculated by summing the modifiable cardiovascula risk components across cardiovascular risk factors not at optimal goal at the time of the encounter, and was calculated for each enrolled patient at the index visit and each subsequent encounter during the intervention period. Annual rate of change in modifiable cardiovascular risk was estimated from all patient encounters. A comparison of the difference in model-estimated rate of change in modifiable cardiovascular risk at 12 months post-index tested the primary efficacy hypothesis.
Time Frame: Index to 12 months post index visit
Population: The patients whose data were included in the primary outcome analysis met eligibility criteria, had an index visit at a randomized clinic at which they were eligible for the Cardiovascular Wizard intervention, and had at least one follow-up visit in a randomized primary care clinic.
Measure: Number; unit: percentage of annual rate of change
Groups:
- Prioritized Clinical Decision Support: Patients and their primary care providers were presented with their patient-specific written advice as to prioritized treatment and lifestyle changes that could reduce their cardiovascular risk, prompted by an electronic health record based alert during their primary care visits.
- Usual Care: Patients and providers were not presented with the prioritized clinical decision support.
Arm/Group | Prioritized Clinical Decision Support | Usual Care
Number analyzed (Participants) | 4550 | 4387
percentage of annual rate of change | 14.2 | 20.8

ADVERSE EVENTS:
Time Frame: The adverse event data was collected on the date of the after-index visit and every subsequent visit through the end of the intervention period on September 19, 2018.
Groups:
- Prioritized Clinical Decision Support: Patients and providers were presented with patient-specific written advice as to prioritized treatment and lifestyle changes that could reduce their cardiovascular risk, prompted by an electronic health record based alert during their primary care visits.
Arm/Group | Prioritized Clinical Decision Support | Usual Care
All-Cause Mortality (participants affected / at risk) | 526/4550 | 581/4837
Serious Adverse Events (participants affected / at risk) | 722/4550 | 763/4387
Other Adverse Events (participants affected / at risk) | 1593/4550 | 1882/4387
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prioritized Clinical Decision Support (N=4550) | Usual Care (N=4387)
In Patient Hospitalization (General disorders) | 702 (1331) | 734 (1415)
Suicide Attempt (General disorders) | 80 (126) | 118 (170)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prioritized Clinical Decision Support (N=4550) | Usual Care (N=4387)
Emergency Room Visit (General disorders) | 1593 (5373) | 1882 (6863)

LIMITATIONS AND CAVEATS:
Because the study was conducted in three large medical groups in the same area of the country, generalizability of results to other care systems or populations is uncertain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-23): https://cdn.clinicaltrials.gov/large-docs/70/NCT02451670/Prot_SAP_000.pdf